CLINICAL TRIAL: NCT00591565
Title: An 8 Week Open-Label Study to Evaluate the Efficacy and Safety of Acamprosate Calcium (Campral) as Augmentation Therapy in Patients With Anxiety Symptoms Who Are Only Partial Responders to SSRI or SNRI Antidepressants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Thomas L. Schwartz, M.D., Assoc Professor, State University of New York - Upstate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMP-MD-15
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Anxiety
Keywords: Anxiety; SSRI; SNRI; Acamprosate
MeSH Terms: conditions — Anxiety Disorders | interventions — Acamprosate

ARMS (1):
- 1 (Experimental): acamprosate tablets
  Interventions: Drug: Acamprosate

INTERVENTIONS:
Drug: Acamprosate — acamprosate 333mg tab, 3 by mouth 3 times a day

SUMMARY:
This study is designed to evaluate anxious patients who are only partially responsive to typical SSRI or SNRI anti-anxiety medication therapy. Patients who are less than 50% anxiety-alleviated on their SSRI medication will be asked to join the study and be placed on Acamprosate as well. This type of add-on therapy is common in outpatient psychiatric care. This is a rater-blinded, patient open-label, non-placebo prospective study, where all subjects will receive Acamprosate for 8 weeks. This study would be the first to date in this treatment-resistant patient population, as the investigators will utilize the a comprehensive set of rating scales in order to best categorize patient responses in regards to anxiety, co-occurring depression, sleep disorders, alcohol use, and social functioning with this drug. This study may be pivotal to the initiation of future double-blind, placebo-controlled studies for this agent

DETAILED DESCRIPTION:
Acamprosate is felt to restore the normal glutamate-GABA balance in the human brain. (Glutamate is a stimulating chemical in the brain, while GABA is an inhibitory chemical in the brain.) This GABA-glutamate balance is felt to play a role in the development of anxiety. Low GABA and high glutamate levels (similar to the state of alcohol withdrawal) are implicated. Symptoms of anxiety may include worry, sweating, nausea, palpitation, tremor, again comparable to that of alcohol withdrawal. Sometimes, GABA-promoting sedative drugs, such as diazepam (Valium) are used to raise GABA activity to ward of anxiety symptoms in the non-alcoholic patient. GABA sedatives are also used to treat alcohol withdrawal to restore balance over the short term. Given the similar glutamate-GABA imbalance in anxiety states and (post)-alcohol withdrawal states, Acamprosate may be a likely candidate to treat anxiety. Acamprosate is now FDA approved to prolong sobriety and decrease alcohol consumption.

The usual initial treatment for anxiety is to use a serotonin neurotransmitter enhancing drug, such as fluoxetine (Prozac). These 'SSRI' drugs, unlike the sedatives noted above, do not have addiction potential and are safer to use. In addition serotonin-norepinephrine facilitating drugs are also used (SNRIs) as alternatives. In the anxiety disorder population, only 30-70% of patient achieve full relief of anxiety symptoms when placed on SSRI monotherapy. The usual second-line choice to promote full anxiety symptom remission is to add a GABA-sedative to the serotonergic SSRI. The authors feel that Acamprosate, given its ability to manipulate the GABA-glutamate balance without major side effects, nor addiction, may be a reasonable add-on or augmentation strategy to better alleviate anxiety in SSRI partial responders.

This study is designed to evaluate anxious patients who are only partially responsive to typical SSRI or SNRI anti-anxiety medication therapy. Patients who are less than 50% anxiety-alleviated on their SSRI medication will be asked to join the study and be placed on Acamprosate as well. This type of add-on therapy is common in outpatient psychiatric care. This is a rater-blinded, patient open-label, non-placebo prospective study, where all subjects will receive Acamprosate for 8 weeks. This study would be the first to date in this treatment-resistant patient population, as the investigators will utilize the a comprehensive set of rating scales in order to best categorize patient responses in regards to anxiety, co-occurring depression, sleep disorders, alcohol use, and social functioning with this drug. This study may be pivotal to the initiation of future double-blind, placebo-controlled studies for this agent

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is obtained.
2. The patient is English-speaking and 18 through 64 years of age inclusive.
3. The patient meets the DSM-IV criteria for anxiety disorder as determined by the MINI and psychiatric evaluation. These include: Post-Traumatic Stress Disorder (PTSD), General Anxiety Disorder (GAD), Social Anxiety, and Panic Disorder.
4. The patient is currently taking a monotherapy SSRI for ≥ 6 weeks and on a stable, adequate therapeutic for ≥ 4 weeks and remains anxiety symptomatic
5. The patient has a total score of at least 16 on the HAM-A scale
6. The patient has a score of at least 7 on the HADS anxiety subscale score at the screening and baseline visits.
7. The patient has a CGI-S rating of 4 or higher at screening
8. The patient is in good health as determined by a medical and psychiatric history, medical examination, and cannot have major medical illness that would jeopardize patient health during the study.
9. Women must be of nonchildbearing potential [i.e., postmenopausal, be surgically sterile (hysterectomy or tubal ligation)] or must meet all of the following conditions: using a reliable, medically accepted form of contraception for at least 60 days before the baseline visit, and agree to continue such use throughout the duration of the study and for 30 days after the final dose of study drug. Reliable forms of contraception include oral, implanted, or injected contraceptives; intrauterine devices in place for at least 3 months; and adequate barrier methods in conjunction with spermicide (abstinence is considered an acceptable contraceptive regimen). Women must be given a pregnancy test (ßHCG), unless they are at least 2 years postmenopausal or surgically sterile, and the results of the test must be negative.
10. The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

1. The patient is on more than one antidepressant or takes a standing sedative anxiolytic
2. The patient has a substance misuse disorder (including alcohol, caffeine, but not nicotine)
3. The patient is a significant risk of suicide
4. The patient has recently started psychotherapy or counseling (within last 6 weeks)
5. The patient has other psychiatric Axis-I disorders as a principal diagnosis (except anxiety) within 6 months of screening and baseline visits; any history of OCD, psychotic disorder, bipolar disorder, or eating disorder, mental retardation, or clear personality disorder. Patient may have a co-morbid substance misuse, depressive or anxiety disorder if it has been in remission for at least 6 months prior to screening visit.
6. The patient has previously participated in any clinical study with acamprosate or treated with acamprosate.
7. The patient has used an investigational drug within 1 month before the screening visit or is participating in a concurrent clinical trial.
8. The patient has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
9. The patient is unlikely to comply with the study protocol, be unreliable in providing ratings, or is unsuitable for any reason, as judged by the investigator.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Schwartz, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University Psychiatry Dept., Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by radio, newspaper and word of mouth
Groups:
- Acamprosate: acamprosate tablets
Period: Overall Study
Arm/Group | Acamprosate
Started | 13
Completed | 8
Not Completed | 5
Not completed — lost follow up, withdrawn | 5

BASELINE CHARACTERISTICS:
Arm/Group | Acamprosate
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at 8 Weeks in the HAM-A Scale
Description: this is a validated clinician administered scale that can range from 0-44 (mild to severe illness).
Time Frame: baseline and 8wk
Population: LOCF if two initial visits were completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acamprosate
Number analyzed (Participants) | 8
units on a scale | 6.12 (1.39)

ADVERSE EVENTS:
Arm/Group | Acamprosate
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acamprosate (N=13)
nausea (Gastrointestinal disorders) | 1 (1)
Vivid Dreams (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
open label design without placebo control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No